CLINICAL TRIAL: NCT04975438
Title: A Phase Ib, Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study of the Clinical Effect, Safety and Tolerability of a Single Intravenous Infusion of GSK1070806 in Moderate to Severe Atopic Dermatitis Patients
Brief Title: Clinical Effect, Safety and Tolerability of GSK1070806 in Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 215253
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Dermatitis, Atopic
Keywords: Eczema activity severity index; GSK1070806
MeSH Terms: conditions — Dermatitis, Atopic | interventions — GSK1070806

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: GSK1070806 (Experimental): Participants received a single dose of 2 mg/kg GSK1070806 as intravenous infusion on Day 1.
  Interventions: Drug: GSK1070806
- Group 1: Placebo (Placebo Comparator): Participants received Placebo as intravenous infusion on Day 1.
  Interventions: Drug: Placebo
- Group 2: Dupilumab-IR with GSK1070806 (Experimental): Participants received a single dose of 2 mg/kg GSK1070806 as intravenous infusion on Day 1.
  Interventions: Drug: GSK1070806
- Group 2: Dupilumab IR with Placebo (Placebo Comparator): Participants received Placebo as intravenous infusion on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK1070806 — GSK1070806 will be administered
  Arms: Group 1: GSK1070806; Group 2: Dupilumab-IR with GSK1070806
Drug: Placebo — Placebo will be administered
  Arms: Group 1: Placebo; Group 2: Dupilumab IR with Placebo

SUMMARY:
This study will evaluate efficacy and safety of GSK1070806 in moderate to severe atopic dermatitis (AtD) participants.

ELIGIBILITY:
Inclusion criteria:

* Moderate to severe AtD (confirmed by a dermatologist) according to the Hannifin and Rajka criteria or Eichenfield revised criteria.
* Onset of AtD symptoms occurring at least 6 months prior to Screening, with stable disease for at least 1 month prior to Screening.
* Eczema Activity Severity Index greater than or equal to (>=)16; Investigator Global Assessment score >=3.
* Group 1- Biologic Naïve: Topical First Line Treatment: Documented recent history (within 6 months before Screening) of: a) either an inadequate response (IR) to out-patient treatment with at least one topical treatment (intermittent topical corticosteroid, topical calcineurin inhibitor), topical inhibitors or Phosphodiesterase 4 inhibitor (Crisaborole); b) or that topical treatments were otherwise not recommended.
* Group 2- Dupilumab-Inadequate Responder: Documented history of an IR to dupilumab: a) either following at least 16 weeks of treatment according to the Investigator's judgement; b) or intolerant to dupilumab owing to adverse events.

Exclusion Criteria:

* Other than AtD, the presence of a significant skin morbidity that will influence the Investigator's ability to assess the severity of the disease (e.g. psoriasis, confirmed or suspected cutaneous T-cell lymphoma, autoimmune bullous disease, fixed drug reaction and Stevens Johnson Syndrome).
* Participants with any uncontrolled medical conditions, other than AtD, that in the opinion of the investigator puts the participant at unacceptable risk or will likely interfere with study assessments or data integrity. Other medical conditions should be stable at the time of screening and be expected to remain stable for the duration of the study.
* Treatment with biologic agents (investigational and marketed monoclonal antibodies) within 12 weeks or 5 pharmacokinetic half-lives (whichever is longer) prior dosing on Day 1.
* Treatment with Janus Activated Kinase inhibitors (e.g. baricitinib, upadacitinib) within 4 weeks or 5 half-lives (whichever is longer) prior to dosing on Day 1.
* Mycophenolate mofetil, azathioprine, methotrexate, or calcineurin inhibitors within 4 weeks of Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2023-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- United States (8):
  - GSK Investigational Site, North Little Rock, Arkansas
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Troy, Michigan
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Sugar Land, Texas
- Canada (2):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, London, Ontario

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 34 participants were enrolled at different centers in Canada and United States.
Pre-assignment Details: The study assessed the impact of GSK1070806 in two groups (Group 1 and Group 2) of participants with moderate-to-severe Atopic Dermatitis (AtD). Group 1 included participants naive to biologic treatment (and who have failed topical therapies) and Group 2 included participants who have not adequately responded (or have been intolerant) to dupilumab (Dupixent).
Groups:
- Group 1: GSK1070806: Participants received a single dose of 2 milligram per kilogram (mg/kg) GSK1070806 as intravenous infusion on Day 1.
- Group 2: Dupilumab- Inadequate Responders (IR) With GSK1070806: Participants received a single dose of 2 mg/kg GSK1070806 as intravenous infusion on Day 1.
Period: Overall Study
Arm/Group | Group 1: GSK1070806 | Group 1: Placebo | Group 2: Dupilumab- Inadequate Responders (IR) With GSK1070806 | Group 2: Dupilumab IR With Placebo
Started | 20 | 10 | 3 | 1
Completed | 18 | 10 | 2 | 1
Not Completed | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population comprised of enrolled analysis set who were assigned to study intervention. Because of the small sample size, summary of baseline/demographics categorical variables are presented as de-identified to prevent risk of participant re-identification.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: GSK1070806 | Group 1: Placebo | Group 2: Dupilumab-IR With GSK1070806 | Group 2: Dupilumab IR With Placebo | Total
Number analyzed (Participants) | 20 | 10 | 3 | 1 | 34
Age, Customized [Count of Participants; unit: Participants]
  De-identified | 20 | 10 | 3 | 1 | 34
Sex/Gender, Customized [Count of Participants; unit: Participants]
  De-identified | 20 | 10 | 3 | 1 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  De-identified | 20 | 10 | 3 | 1 | 34

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline (PCFB) in Eczema Area and Severity Index (EASI) Score at Week 12 in Group 1
Description: EASI scoring system is standardized clinical tool for assessment of extent (area) and severity of atopic dermatitis (AD). Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk and lower limbs on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % body surface area with AD in body region: 0 (0%), 1=1-9%; 2=10-29%; 3=30-49%; 4=50-69%; 5=70-89%; 6=90-100% The final EASI score was obtained by weight-averaging these 4 scores and scores ranged from 0 to 72, with higher scores= more severe or extensive condition. Posterior Median presented from Bayesian analysis under the hypothetical strategy. The percent change from baseline in the EASI score at week 12 in group 1 is reported here. Data reported as 'Median' refers to 'Posterior Median' and '95% Confidence Interval' refers to '95% Credible Interval'.
Time Frame: Baseline (Day 1) and at Week 12
Population: The Safety Set included all randomized participants who received the study intervention. Participants were analyzed according to the intervention they actually received. Number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Percent Change
Groups:
- Group 1: GSK1070806: In group 1, participants received a single dose of GSK1070806 2 mg/kg intravenous infusion on Day 1.
- Group 1: Placebo: In group 1, participants received Placebo intravenous infusion on Day 1.
Arm/Group | Group 1: GSK1070806 | Group 1: Placebo
Number analyzed (Participants) | 19 | 9
Percent Change | -66.11 [-78.65 to -53.54] | -32.81 [-46.59 to -20.34]
Statistical Analysis 1: Comparison: Group 1: GSK1070806 vs Group 1: Placebo; Test type: Other; Posterior Median Difference = -33.21, 95% CI 2-sided [-50.96 to -14.84] — The posterior median of the difference (GSK1070806 - placebo) and 95% credible interval in PCFB in the EASI is presented. Analysis was performed using Bayesian analysis under the hypothetical strategy using an informative prior (robust MAP prior)

2. Secondary Outcome: Change From Baseline in EASI Score at Week 12 in Group 1
Description: EASI scoring system is standardized clinical tool for assessment of extent (area) and severity of atopic dermatitis (AD). Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk and lower limbs on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % body surface area with AD in body region: 0 (0%), 1=1-9%; 2=10-29%; 3=30-49%; 4=50-69%; 5=70-89%; 6=90-100% The final EASI score was obtained by weight-averaging these 4 scores and scores ranged from 0 to 72, with higher scores= more severe or extensive condition. Posterior Median presented from Bayesian analysis under the hypothetical strategy. The change from baseline in the EASI score at week 12 in group 1 is reported here. Data reported as 'Median' refers to 'Posterior Median' and '95% Confidence Interval' refers to '95% Credible Interval'.
Time Frame: Baseline (Day 1) and at Week 12
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Group 1: GSK1070806 | Group 1: Placebo
Number analyzed (Participants) | 19 | 9
Scores on a Scale | -16.83 [-20.30 to -13.36] | -7.15 [-12.12 to -2.20]
Statistical Analysis 1: Comparison: Group 1: GSK1070806 vs Group 1: Placebo; Test type: Other; Posterior Median Difference = -9.68, 95% CI 2-sided [-15.70 to -3.60] — The posterior median of the difference (GSK1070806 - placebo) and 95% credible interval in PCFB in the EASI is presented. Analysis was performed using Bayesian analysis with vague priors and adjusting for baseline EASI

3. Secondary Outcome: Number of Participants Achieving EASI-50, ≥ 50% Reduction in EASI Score at Week 12 in Group 1
Description: EASI scoring system is standardized clinical tool for assessment of extent (area) and severity of atopic dermatitis (AD). Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk and lower limbs on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % body surface area with AD in body region: 0 (0%), 1=1-9%; 2=10-29%; 3=30-49%; 4=50-69%; 5=70-89%; 6=90-100% The final EASI score was obtained by weight-averaging these 4 scores and scores ranged from 0 to 72, with higher scores= more severe or extensive condition. The EASI-50 responder is defined as a participant who achieves a ≥ 50% improvement from baseline in the EASI score.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: GSK1070806 | Group 1: Placebo
Number analyzed (Participants) | 19 | 9
Participants
  Responder | 14 | 3
  Non-responder | 5 | 6

4. Secondary Outcome: Number of Participants Achieving EASI-75, ≥ 75% Reduction in EASI Score at Week 12 in Group 1
Description: EASI scoring system is standardized clinical tool for assessment of extent (area) and severity of atopic dermatitis (AD). Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk and lower limbs on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % body surface area with AD in body region: 0 (0%), 1=1-9%; 2=10-29%; 3=30-49%; 4=50-69%; 5=70-89%; 6=90-100% The final EASI score was obtained by weight-averaging these 4 scores and scores ranged from 0 to 72, with higher scores= more severe or extensive condition. The EASI-75 responder is defined as a participant who achieves a ≥ 75% improvement from baseline in the EASI score.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: GSK1070806 | Group 1: Placebo
Number analyzed (Participants) | 19 | 9
Participants
  Responder | 7 | 1
  Non-responder | 12 | 8

5. Secondary Outcome: Number of Participants Achieving EASI-90, ≥ 90% Reduction in EASI Score at Week 12 in Group 1
Description: EASI scoring system is standardized clinical tool for assessment of extent (area) and severity of atopic dermatitis (AD). Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk and lower limbs on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % body surface area with AD in body region: 0 (0%), 1=1-9%; 2=10-29%; 3=30-49%; 4=50-69%; 5=70-89%; 6=90-100% The final EASI score was obtained by weight-averaging these 4 scores and scores ranged from 0 to 72, with higher scores= more severe or extensive condition. The EASI-90 responder is defined as a participant who achieves a ≥ 90% improvement from baseline in the EASI score.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: GSK1070806 | Group 1: Placebo
Number analyzed (Participants) | 19 | 9
Participants
  Responder | 5 | 1
  Non-responder | 14 | 8

6. Secondary Outcome: Number of Participants With Investigator Global Assessment (IGA) Score of 0 or 1 at Week 12 in Group 1
Description: The Investigator Global Assessment (IGA) is a clinical tool for assessing the current state/severity of a participant's atopic dermatitis. It is a static 5-point morphological assessment of overall disease severity determined by the investigator, sub-investigator, or trained healthcare professional with required qualifications on a scale of 0 to 4 where, 0-clear, 1-almost clear, 2-mild, 3-moderate, and 4- severe. Higher score indicates severity of disease. A Responder is defined as a participant who had an IGA score of 0 or 1 at each visit.
Time Frame: At Week 12
Population: The analysis was performed on Safety Set that included all randomized participants who received the study intervention. Participants were analyzed according to the intervention they actually received. Number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: GSK1070806 | Group 1: Placebo
Number analyzed (Participants) | 19 | 9
Participants
  Almost Clear (1) | 4 | 1
  Clear (0) | 1 | 0

7. Secondary Outcome: Percent Change From Baseline in EASI Score at Week 12 in Group 2
Description: EASI scoring system is standardized clinical tool for assessment of extent (area) and severity of atopic dermatitis (AD). Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk and lower limbs on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % body surface area with AD in body region: 0 (0%), 1=1-9%; 2=10-29%; 3=30-49%; 4=50-69%; 5=70-89%; 6=90-100% The final EASI score was obtained by weight-averaging these 4 scores and scores ranged from 0 to 72, with higher scores= more severe or extensive condition. NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation (SD) was not derived.
Time Frame: Baseline (Day 1) and at Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- Group 2: Dupilumab-Inadequate Responders (IR) With GSK1070806: In group 2, participants received a single dose of GSK1070806 of 2 mg/kg intravenous infusion on Day 1.
- Group 2: Dupilumab IR With Placebo: In group 2, participants received Placebo intravenous infusion on Day 1.
Arm/Group | Group 2: Dupilumab-Inadequate Responders (IR) With GSK1070806 | Group 2: Dupilumab IR With Placebo
Number analyzed (Participants) | 3 | 1
Percent Change | -94.213 (8.1841) | -38.868 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived.

8. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) - Groups 1 and 2
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. SAEs are defined as any serious adverse event that, at any dose which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect and other situations as per investigator's medical or scientific judgment.
Time Frame: Up to Week 24
Population: The analysis was performed on the Safety Set that included all randomized participants who received the study intervention. Participants were analyzed according to the intervention they actually received. Number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1 and 2: GSK1070806: Participants received a single dose of 2 mg/kg of GSK1070806 intravenous infusion in Group 1 and 2.
- Group 1 and 2: Placebo: Participants received Placebo intravenous infusion in Group 1 and 2.
Arm/Group | Group 1 and 2: GSK1070806 | Group 1 and 2: Placebo
Number analyzed (Participants) | 23 | 11
Participants
  Adverse Events | 10 | 6
  Serious Adverse Events | 0 | 0

9. Secondary Outcome: Number of Participants With Worst Case Vital Signs Results by Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline - Groups 1 and 2
Description: Vital signs included diastolic blood pressure (DBP), systolic blood pressure (SBP), pulse rate (PR) and body temperature were measured after resting for at least 5 minutes in semi-supine position. PCI ranges- SBP (millimeters of mercury[mmHg]): <85 (low) or >160 (high), DBP (mmHg): <45 (low) or >100 (high), PR (beats per minute): <40 (low) or >110 (high) and body temperature (degrees Celsius) <=35.5 (low) or >38.0 (high). Participants with worst case results relative to PCI criteria and who had values "to high" are reported here. Participants with a missing baseline value are assumed to have a within range value.
Time Frame: Up to Week 24
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 and 2: GSK1070806 | Group 1 and 2: Placebo
Number analyzed (Participants) | 23 | 11
Participants
  Diastolic Blood Pressure (mmHg), Worst Case Post-Baseline,To Low | 0 | 0
  Diastolic Blood Pressure (mmHg),Worst Case Post-Baseline, To w/in Range or No Change | 22 | 10
  Diastolic Blood Pressure (mmHg),Worst Case Post-Baseline, To High | 1 | 1
  Pulse Rate (beats/min),Worst Case Post-Baseline,To Low | 0 | 0
  Pulse Rate (beats/min),Worst Case Post-Baseline, To w/in Range or No Change | 23 | 11
  Pulse Rate (beats/min),Worst Case Post-Baseline, To High | 0 | 0
  Systolic Blood Pressure (mmHg),Worst Case Post-Baseline,To Low | 0 | 0
  Systolic Blood Pressure (mmHg),Worst Case Post-Baseline, To w/in Range or No Change | 22 | 11
  Systolic Blood Pressure (mmHg),Worst Case Post-Baseline, To High | 1 | 0
  Temperature (C),Worst Case Post-Baseline,To Low | 1 | 0
  Temperature (C),Worst Case Post-Baseline, To w/in Range or No Change | 22 | 11
  Temperature (C), Worst Case Post-Baseline, To High | 0 | 0

10. Secondary Outcome: Number of Participants With Worst Case 12-lead Electrocardiogram (ECG) Post-Baseline Relative to Baseline - Groups 1 and 2
Description: Twelve lead ECG was obtained using an ECG machine that automatically calculated the heart rate and measured QTc, PR, QRS intervals. Participants with clinically significant changes relative to baseline are reported here. Clinically significant findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Up to Week 24
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 and 2: GSK1070806 | Group 1 and 2: Placebo
Number analyzed (Participants) | 21 | 10
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Worst Case Urinalysis Results Post-Baseline Relative to Baseline - Groups 1 and 2
Description: Urine samples were collected to assess urine glucose, bilirubin, protein, occult blood, Leukocyte Esterase and ketones using dipstick method. Participants with clinically significant changes relative to baseline are reported here. Clinically significant findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Baseline was defined as the latest pre-dose assessment.
Time Frame: Up to Week 24
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 and 2: GSK1070806 | Group 1 and 2: Placebo
Number analyzed (Participants) | 22 | 11
Participants | 0 | 0

12. Secondary Outcome: Number of Participants With Worst Case Chemistry Results by Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline - Groups 1 and 2
Description: Blood samples were collected for analysis of chemistry parameters. PCI ranges were >3*Upper limit of normal (ULN) units per liter (U/L)(Alanine Aminotransferase [ALT]), >3*ULN (U/L) (Aspartate Aminotransferase ([AST]), >2*ULN (Alkaline Phosphatase [ALP]) (U/L), >2*ULN (micromoles per liter) (bilirubin), <3 or >6.5 mmol/L (potassium), <130 or >160 mmol/L (sodium), <1.5 or >3.25 mmol/L (Corrected Calcium) and >40 mmol/L (Urea). Participants with worst case results relative to PCI criteria and who had values "to high" are reported here. Participants with a missing baseline value are assumed to have a within range value.
Time Frame: Up to Week 24
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 and 2: GSK1070806 | Group 1 and 2: Placebo
Number analyzed (Participants) | 23 | 11
Participants
  Alanine Aminotransferase (IU/L),Worst Case Post-Baseline,To Low | 0 | 0
  Alanine Aminotransferase (IU/L),Worst Case Post-Baseline,To W/in Range or No Change | 22 | 11
  Alanine Aminotransferase (IU/L),Worst Case Post-Baseline,To High | 1 | 0
  Albumin (g/L),Worst Case Post-Baseline,To Low | 0 | 0
  Albumin (g/L),Worst Case Post-Baseline,To W/in Range or No Change | 23 | 11
  Albumin (g/L),Worst Case Post-Baseline,,To High | 0 | 0
  Alkaline Phosphatase (IU/L),Worst Case Post-Baseline,To Low | 0 | 0
  Alkaline Phosphatase (IU/L),Worst Case Post-Baseline,To W/in Range or No Change | 23 | 11
  Alkaline Phosphatase (IU/L),Worst Case Post-Baseline,,To High | 0 | 0
  Aspartate Aminotransferase (IU/L),Worst Case Post-Baseline,To Low | 0 | 0
  Aspartate Aminotransferase (IU/L),Worst Case Post-Baseline,To W/in Range or No Change | 22 | 10
  Aspartate Aminotransferase (IU/L),Worst Case Post-Baseline,,To High | 1 | 1
  Bilirubin (umol/L),Worst Case Post-Baseline,To Low | 0 | 0
  Bilirubin (umol/L),Worst Case Post-Baseline,To W/in Range or No Change | 0 | 0
  Bilirubin (umol/L),Worst Case Post-Baseline,To High | 23 | 11
  Calcium Corrected for Albumin (mmol/L),Worst Case Post-Baseline,To Low | 0 | 0
  Calcium Corrected for Albumin (mmol/L),Worst Case Post-Baseline,To W/in Range or No Change | 23 | 11
  Calcium Corrected for Albumin (mmol/L),Worst Case Post-Baseline,To High | 0 | 0
  Potassium (mmol/L),Worst Case Post-Baseline,To Low | 0 | 0
  Potassium (mmol/L),Worst Case Post-Baseline,To W/in Range or No Change | 23 | 11
  Potassium (mmol/L),Worst Case Post-Baseline,To High | 0 | 0
  Sodium (mmol/L),Worst Case Post-Baseline,To Low | 2 | 0
  Sodium (mmol/L),Worst Case Post-Baseline,To W/in Range or No Change | 21 | 11
  Sodium (mmol/L),Worst Case Post-Baseline,To High | 0 | 0
  Urea (mmol/L),Worst Case Post-Baseline,To Low | 0 | 0
  Urea (mmol/L),Worst Case Post-Baseline,To W/in Range or No Change | 23 | 11
  Urea (mmol/L),Worst Case Post-Baseline,To High | 0 | 0

13. Secondary Outcome: Number of Participants With Worst Case Hematology Results by Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline - Groups 1 and 2
Description: Blood samples were collected for analysis of hematology parameters. The ranges for the hematology parameters are as follows: Hematocrit [High >0.54 Proportion of red blood cells in blood, Low <0.1 Proportion of red blood cells in blood], Haemoglobin [Higher: > 185 grams/Litre (g/L) Low: less than (<) 100 g/L ], Lymphocytes [<0.8 10^9/L], Neutrophils [<1.5 10^9/L], Platelets [High: > 999 10^9/ L and Low: < 100 10^9/ L] and White blood cells [Low:<2 10^9/L]. Participants were counted in worst case category that their value changes to (low, within range or no change or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (for example [e.g.], High to High), or whose value became within range, were recorded in "To within Range or No Change" category. Participants were counted twice if participant has values that changed 'To Low' & 'To High', so the percentages may not add to 100%.
Time Frame: Up to Week 25
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 and 2: GSK1070806 | Group 1 and 2: Placebo
Number analyzed (Participants) | 23 | 11
Participants
  Hematocrit (fraction of 1),Worst Case Post-Baseline,To Low | 0 | 0
  Hematocrit (fraction of 1),Worst Case Post-Baseline,To W/in Range or No Change | 22 | 11
  Hematocrit (fraction of 1),Worst Case Post-Baseline,To High | 1 | 0
  Hemoglobin (g/L),Worst Case Post-Baseline,To Low | 2 | 0
  Hemoglobin (g/L),Worst Case Post-Baseline,To W/in Range or No Change | 21 | 11
  Hemoglobin (g/L),Worst Case Post-Baseline,To High | 0 | 0
  Leukocytes (10^9/L),Worst Case Post-Baseline,To Low | 0 | 0
  Leukocytes (10^9/L),Worst Case Post-Baseline,To W/in Range or No Change | 23 | 11
  Leukocytes (10^9/L),Worst Case Post-Baseline,To High | 0 | 0
  Lymphocytes (10^9/L),Worst Case Post-Baseline,To Low | 2 | 2
  Lymphocytes (10^9/L),Worst Case Post-Baseline,To W/in Range or No Change | 21 | 9
  Lymphocytes (10^9/L),Worst Case Post-Baseline,To High | 0 | 0
  Neutrophils (10^9/L),Worst Case Post-Baseline,To Low | 2 | 0
  Neutrophils (10^9/L),Worst Case Post-Baseline,To W/in Range or No Change | 21 | 11
  Neutrophils (10^9/L),Worst Case Post-Baseline,To High | 0 | 0
  Platelets (10^9/L),Worst Case Post-Baseline,To Low | 0 | 0
  Platelets (10^9/L),Worst Case Post-Baseline,To W/in Range or No Change | 23 | 11
  Platelets (10^9/L),Worst Case Post-Baseline,To High | 0 | 0

14. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA)- Groups 1 and 2
Description: Serum samples were analyzed for the presence of antibodies using a validated assay method. The treatment emergent ADA assay results up to week 24 are reported.
Time Frame: Up to Week 24
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 and 2: GSK1070806 | Group 1 and 2: Placebo
Number analyzed (Participants) | 22 | 11
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 and up to Week 24
Description: Safety Set comprised of all randomized participants who received study intervention and reported for both Group 1 and group 2 combined as pre-specified in the protocol objectives.
Groups:
- GSK1070806: Group-1, Biologic naive and group-2, Dupilumab-Inadequate (Dupi-IR) Responder participants received a single dose of 2 mg/kg of GSK1070806 intravenous infusion on Day 1
- Placebo: Participants received Placebo intravenous infusion in group 1 and 2 on Day 1.
Arm/Group | GSK1070806 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/11
Other Adverse Events (participants affected / at risk) | 10/23 | 6/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1070806 (N=23) | Placebo (N=11)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Neutrophil count abnormal (Investigations) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
White blood cell disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT04975438/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT04975438/SAP_001.pdf